CLINICAL TRIAL: NCT04034719
Title: Benefit of Scarf Support on Skin-to-skin Time and Portage in Neonatology and at Home(PAPSE)
Brief Title: Benefit of Scarf Support on Skin-to-skin Time and Portage in Neonatology and at Home
Acronym: PAPSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19CH089; 2019-A01113-54 (Other: ANSM)
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-01

CONDITIONS: Infant, Newborn, Disease
Keywords: Newborn; Parents; Carrying; Skin-to-skin; Scarf
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Newborn hospitalized in the neonatal department with their parent will be included.
  They will have a portage scarf to help them to keep their child skin-to-skin
  Interventions: Other: portage scarf
- Control group (Active Comparator): Newborn hospitalized in the neonatal department with their parent will be included.
  They wont have a portage scarf.
  Interventions: Other: usual practice

INTERVENTIONS:
Other: portage scarf — Parents will be carried their newborn with the portage scarf provided by the department.
  Arms: Experimental group
Other: usual practice — Parents will be carried their newborn as their usual practice.
  Arms: Control group

SUMMARY:
Carrying (or kangaroo carrying) is known to reduce neonatal and child morbidity and mortality and improves the quality of survival of premature and term children during the most fragile growth period, the first thousand days of life. Carrying is also a growing brain protection technique and becomes a routine of care in all neonatal units around the world.

In University hospital of Saint-Etienne, the developmental care program has been developed since 2002 in all neonatology units and advocates the practice of skin-to-skin carrying between the parent (father or mother) and his baby, from the time of the hospitalization. Professionals in units who have long been thinking about the concept of attachment and the benefits of skin-to-skin, wish to validate the use of the wearing scarf as a tool for the practice of skin -in-skin in neonatology then back home by performing a randomized monocentric prospective longitudinal study.

DETAILED DESCRIPTION:
This study it's a single-center, prospective, randomized study to evaluate the benefit of the scarf in the practice of skin-to-skin and portage (PAPSE Group) compared to a Skin-to-Skin and Carry Without Scarf (PAP group).

ELIGIBILITY:
Inclusion Criteria:

For the child:

* Any newborn regardless of gestational age and postnatal age hospitalized in the neonatology department of the University Hospital of Saint-Etienne

For the parent (father or mother):

* Be a parent of a child eligible for the research protocol

Exclusion Criteria:

For the child:

* Need for sedation or analgesia for the duration of the study
* Orthopedic pathology incompatible with the practice of carrying
* Other medical contraindications to carriage
* Absence of parents

For the parent (father or mother):

* Family, social or psychological situation compromising the evaluation
* No fluency in the French language

Max Age: 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Number of minuts with portage skin-to-skin | From inclusion to 2 months after exit
  Measured in minutes by the time sheet of presence.

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No